CLINICAL TRIAL: NCT04798222
Title: An Open-label, Randomized, Parallel Group, Four/Five Period, Eight Treatment Cross-over, Single Oral Dose Study to Assess the Relative Bioavailability of Different Formulations of AZD9977 and Dapagliflozin and Influence of Food in Selected Formulations in Healthy Volunteers
Brief Title: Study to Assess the Bioavailability of Different Formulations of AZD9977 and Dapagliflozin and Influence of Food in Selected Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D6402C00003; 2021-000483-30 (EudraCT Number)
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure
Keywords: Bioavailability; Oral selective mineralocorticoid receptor modulator; Pharmacokinetics; Dapagliflozin; AZD9977
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Group 1: Treatment Sequence ABECD (Experimental): Participants will receive a single oral dose of Treatments A, B, E, C, and D in Treatment periods 1 to 5 on Day 1 of the study.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D; Drug: Treatment E
- Group 1: Treatment Sequence BACED (Experimental): Participants will receive a single oral dose of Treatments B, A, C, E, and D in Treatment periods 1 to 5 on Day 1 of the study.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D; Drug: Treatment E
- Group 1: Treatment Sequence CDBEA (Experimental): Participants will receive a single oral dose of Treatments C, D, B, E, and A in Treatment periods 1 to 5 on Day 1 of the study.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D; Drug: Treatment E
- Group 1: Treatment Sequence EADBC (Experimental): Participants will receive a single oral dose of Treatments E, A, D, B, and C in Treatment periods 1 to 5 on Day 1 of the study.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D; Drug: Treatment E
- Group 2: Treatment Sequence AFHG (Experimental): Participants will receive a single oral dose of Treatments A, F, H, and G in Treatment periods 1 to 4 on Day 1 of the study.
  Interventions: Drug: Treatment A; Drug: Treatment F; Drug: Treatment G; Drug: Treatment H
- Group 2: Treatment Sequence FGAH (Experimental): Participants will receive a single oral dose of Treatments F, G, A, and H in Treatment periods 1 to 4 on Day 1 of the study.
  Interventions: Drug: Treatment A; Drug: Treatment F; Drug: Treatment G; Drug: Treatment H
- Group 2: Treatment Sequence GHFA (Experimental): Participants will receive a single oral dose of Treatments G, H, F, and A in Treatment periods 1 to 4 on Day 1 of the study.
  Interventions: Drug: Treatment A; Drug: Treatment F; Drug: Treatment G; Drug: Treatment H
- Group 2: Treatment Sequence HAGF (Experimental): Participants will receive a single oral dose of Treatments H, A, G, and F in Treatment periods 1 to 4 on Day 1 of the study.
  Interventions: Drug: Treatment A; Drug: Treatment F; Drug: Treatment G; Drug: Treatment H

INTERVENTIONS:
Drug: Treatment A — Participants will receive oral AZD9977 Dose A capsule and 10 mg dapagliflozin tablet in fasted condition.
Drug: Treatment B — Participants will receive oral AZD9977 Dose A capsule and 10 mg dapagliflozin capsule 1 in fasted condition.
  Arms: Group 1: Treatment Sequence ABECD; Group 1: Treatment Sequence BACED; Group 1: Treatment Sequence CDBEA; Group 1: Treatment Sequence EADBC
Drug: Treatment C — Participants will receive oral AZD9977 Dose A capsule and 10 mg dapagliflozin capsule 1 in fed condition
  Arms: Group 1: Treatment Sequence ABECD; Group 1: Treatment Sequence BACED; Group 1: Treatment Sequence CDBEA; Group 1: Treatment Sequence EADBC
Drug: Treatment D — Participants will receive oral AZD9977 Dose A capsule and 10 mg dapagliflozin capsule 2 in fasted condition.
  Arms: Group 1: Treatment Sequence ABECD; Group 1: Treatment Sequence BACED; Group 1: Treatment Sequence CDBEA; Group 1: Treatment Sequence EADBC
Drug: Treatment E — Participants will receive oral AZD9977 Dose A capsule and 10 mg dapagliflozin capsule 2 in fed condition.
  Arms: Group 1: Treatment Sequence ABECD; Group 1: Treatment Sequence BACED; Group 1: Treatment Sequence CDBEA; Group 1: Treatment Sequence EADBC
Drug: Treatment F — Participants will receive oral AZD9977 Dose A capsule and 10 mg dapagliflozin capsule 3 in fasted condition.
  Arms: Group 2: Treatment Sequence AFHG; Group 2: Treatment Sequence FGAH; Group 2: Treatment Sequence GHFA; Group 2: Treatment Sequence HAGF
Drug: Treatment G — Participants will receive oral AZD9977 Dose A capsule and 10 mg dapagliflozin capsule 4 in fasted condition.
  Arms: Group 2: Treatment Sequence AFHG; Group 2: Treatment Sequence FGAH; Group 2: Treatment Sequence GHFA; Group 2: Treatment Sequence HAGF
Drug: Treatment H — Participants will receive oral dose of dapagliflozin capsule in fasted condition.
  Arms: Group 2: Treatment Sequence AFHG; Group 2: Treatment Sequence FGAH; Group 2: Treatment Sequence GHFA; Group 2: Treatment Sequence HAGF

SUMMARY:
The primary purpose of the study is to evaluate relative bioavailability of AZD9977 and dapagliflozin and compare the plasma concentration time profiles after dosing with different capsule formulations containing both AZD9977 and dapagliflozin or solely dapagliflozin, the AZD9977 capsule, and dapagliflozin tablet under fasted conditions.

DETAILED DESCRIPTION:
The study will be conducted at 2 study centers in Germany.

Eligible participants will be randomized to one of the 8 treatment sequences (4 unique sequences to Group 1 and 4 unique sequences to Group 2). In Group 1, participants will receive 5 single dose treatments, while in Group 2 participants will receive 4 single dose treatments.

Below treatments A, B, C, D and E will be given to participants in Group 1 and treatments A, F, G and H will be given to participants in Group 2 in randomized order:

1. Treatment A: AZD9977 Dose A + 10 mg dapagliflozin tablet, fasted
2. Treatment B: AZD9977 Dose A + 10 mg dapagliflozin capsule 1, fasted
3. Treatment C: AZD9977 Dose A + 10 mg dapagliflozin capsule 1, fed
4. Treatment D: AZD9977 Dose A + 10 mg dapagliflozin capsule 2, fasted
5. Treatment E: AZD9977 Dose A + 10 mg dapagliflozin capsule 2, fed
6. Treatment F: AZD9977 Dose A + 10 mg dapagliflozin capsule 3, fasted
7. Treatment G: AZD9977 Dose A + 10 mg dapagliflozin capsule 4, fasted
8. Treatment H: 10 mg dapagliflozin capsule, fasted

The study will comprise of the following:

* A screening period of maximum 21 days.
* Four or five treatment periods during which participants will be resident at the study center from the day before dosing until at least 72 hours after the final dose.
* A final visit within 5 to 7 days after administration of the last treatment.

Each participant will receive single dose treatments under fasted or fed conditions, separated by at least 4 days washout.

Each participant will be involved in the study for approximately 6 to 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants of non-childbearing potential with suitable veins for cannulation or repeated venipuncture at screening
* Females must have a negative pregnancy test at the screening Visit and a negative urine pregnancy test at admission to the study center, must not be lactating and must be of non childbearing potential
* Have a body mass index between 18 and 29.9 kg/m^2, inclusive, and weigh at least 50 kg and no more than 100 kg, inclusive, at screening

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results at screening, as judged by the Investigator
* Any clinically significant abnormal findings in vital signs, and 12-lead electrocardiogram as judged by the Investigator
* Any positive result on screening for serum hepatitis B surface antigen or anti-hemoglobin antibody, hepatitis C antibody, and human immunodeficiency virus antibody
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months (or 5 half lives, whichever is longer) of the first administration of IMP in this study
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity or history of hypersensitivity to drugs with a similar chemical structure or class to AZD9977 or dapagliflozin
* Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the 3 months prior to screening
* Participant has a positive test result for Severe acute respiratory syndrome coronavirus 2 reverse transcriptase polymerase chain reaction at admission
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP
* Use of any prescribed or non prescribed medication including antacids, analgesics, hormone replacement therapy, herbal remedies, megadose vitamins and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half life
* Participants who have previously received AZD9977 or dapagliflozin
* Judgment by the Investigators that the participant should not participate in the study if they have any ongoing or recent minor medical complaints
* Participants who cannot communicate reliably with the Investigator and/or is not able to read, speak and understand the German language
* Participant has clinical signs and symptoms consistent with corona virus disease 2019 (COVID-19), or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on first admission
* History of severe COVID-19 infection (hospitalization, extracorporeal membrane oxygenation, mechanically ventilated) as judged by the Investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of AUCinf of AZD9977 and dapagliflozin, after dosing with different capsule formulations containing both AZD9977 and dapagliflozin or solely dapagliflozin, the AZD9977 capsule, and dapagliflozin tablet under fasted conditions.
Area under the plasma concentration time curve from zero to the last quantifiable concentration (AUClast) | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of AUClast of AZD9977 and dapagliflozin, after dosing with different capsule formulations containing both AZD9977 and dapagliflozin or solely dapagliflozin, the AZD9977 capsule, and dapagliflozin tablet under fasted conditions.
Maximum observed plasma (peak) drug concentration (Cmax) | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of Cmax of AZD9977 and dapagliflozin, after dosing with different capsule formulations containing both AZD9977 and dapagliflozin or solely dapagliflozin, the AZD9977 capsule, and dapagliflozin tablet under fasted conditions.
Drug concentration in plasma at 24 hours post-dose (C24) | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of C24 of AZD9977 and dapagliflozin, after dosing with different capsule formulations containing both AZD9977 and dapagliflozin or solely dapagliflozin, the AZD9977 capsule, and dapagliflozin tablet under fasted conditions.

SECONDARY OUTCOMES:
AUCinf of AZD9977 and dapagliflozin | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of AUCinf of AZD9977 and dapagliflozin after dosing with 2 different capsule formulations (AZD9977 + dapagliflozin) under fed and fasted conditions.
AUClast of AZD9977 and dapagliflozin | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of AUClast of AZD9977 and dapagliflozin after dosing with 2 different capsule formulations (AZD9977 + dapagliflozin) under fed and fasted conditions.
Cmax of AZD9977 and dapagliflozin | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of Cmax of AZD9977 and dapagliflozin after dosing with 2 different capsule formulations (AZD9977 + dapagliflozin) under fed and fasted conditions.
C24 of AZD9977 and dapagliflozin | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of C24 of AZD9977 and dapagliflozin after dosing with 2 different capsule formulations (AZD9977 + dapagliflozin) under fed and fasted conditions.
AUCinf of AZD9977 | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of AUCinf of AZD9977 in different capsules against each other under fasted conditions.
AUClast of AZD9977 | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of AUClast of AZD9977 in different capsules against each other under fasted conditions.
Cmax of AZD9977 | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of Cmax of AZD9977 in different capsules against each other under fasted conditions.
C24 of AZD9977 | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of C24 of AZD9977 in different capsules against each other under fasted conditions.
AUCinf of dapagliflozin | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of AUCinf of dapagliflozin in different capsules against each other under fasted conditions.
AUClast of dapagliflozin | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of AUClast of dapagliflozin in different capsules against each other under fasted conditions.
Cmax of dapagliflozin | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of Cmax of dapagliflozin in different capsules against each other under fasted conditions.
C24 of dapagliflozin | Day 1 until Day 4 of each Treatment Period (Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
  Evaluation of C24 of dapagliflozin in different capsules against each other under fasted conditions.
Number of participants with adverse events | From screening until follow-up visit (5 to 7 days post final dose)
  Assessment of the safety and tolerability of single doses of AZD9977 and dapagliflozin in healthy participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ozan Dursun, Principal Investigator — Parexel Early Phase Clinical Unit Berlin Campus DRK Kliniken Berlin Westend, Haus 31 Spandauer Damm 130 14050 Berlin Germany; Alen Jambrecina, Principal Investigator — CTC North GmbH & Co. KG Martinistrasse 64 20251 Hamburg Germany
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home